CLINICAL TRIAL: NCT04751760
Title: Feasibility Study of a New Immunoglobulin E (IgE) Assay Method in Urine and Blood
Brief Title: Feasibility Study of a New Immunoglobulin E (IgE) Assay Method
Acronym: LuLISA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/20/0293
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Allergy and Immunology
Keywords: IgE assay; food allergy/ hypersensitivity; respiratory allergy/ hypersensitivity; hymenopter allergy/ hypersensitivity
MeSH Terms: conditions — Hypersensitivity | interventions — Urination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People with sensitization or allergy: blood and urine will be collected during a blood test scheduled for the follow-up of the patient
  Interventions: Biological: collection of blood and urine

INTERVENTIONS:
Biological: collection of blood and urine — blood and urine will be collected during a blood test scheduled for the follow-up of the patient

SUMMARY:
The main objective is to study the feasibility of a new specific IgE assay using a bioluminescence technique in a pediatric and adult allergic population. For this, we will collect blood, and urine during a blood test scheduled for the follow-up of the patient.

DETAILED DESCRIPTION:
Allergy is a raising public health problem. Specific IgE assays are useful tools to investigate the physiopathology of allergies. This method is achieved mainly by the ImmunoCAP enzyme immunoassay technique. This is an expensive test that requires a significant amount of blood. This is a limitation particularly in children. The time to get the results is long and a second consultation has to be scheduled in order to communicate the results to the patients. The main objective of this study is to assess the feasibility of a new specific IgE assay, named LuLISA, using a bioluminescence technique in urine and blood samples from pediatric and adult allergic population. This technique was recently published for the quantification of IgE against two peanut allergens and needs to be extended for the detection of other major allergens. A secondary objective is the evaluation of the time needed to obtain results.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 6 months' old or older
* Sensitization or allergy towards a trophallergen, an aeroallergen, hymenoptera venom or drug proven by:

  * positive skin test (s)
  * and / or IgE specific (s)> 0.1 kUA / L
  * and / or anamnesis in favor of an allergic reaction of mediated IgE
* Social coverage up to date

Exclusion Criteria:

* Children younger than 6 months'old
* Children's weight less than 10 kg
* Pregnant or breastfeeding women
* Patients with cystic fibrosis
* Patients with dysimmune or autoimmune pathology
* Anamnesis in favor of a delayed allergy or a contact allergy.

Ages: 6 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients followed at the Toulouse University Hospital and presenting sensitization or allergy towards a trophallergen, an aeroallergen, hymenoptera venom or drug
Sampling Method: Probability Sample
Enrollment: 1376 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
Estimation of the the correlation of specific IgE concentrations for a given allergen analyzed using two different methods | Day 0
  specific IgE concentrations for a given allergen will be measured by both LuLISA and ImmunoCAP and the results will be compared

SECONDARY OUTCOMES:
To study the correlation between the results of specific serum and urinary IgE dosages by LuLISA | Day 0
  specific IgE concentrations for a given allergen will be measured in the sera and the urine from the same patient and the results will be compared
To study the correlation between the results of specific IgE dosages in the venous blood and the capillary blood | Day 0
  specific IgE concentrations for a given allergen will be measured in the venous blood and the capillary blood from the same patient and the results will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Marine Michelet, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - University Hospital, Toulouse
  - Larrey hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No